CLINICAL TRIAL: NCT02856321
Title: PerLE (Peroneus Longus Evaluation): A Study Evaluating the Efficacy of Injection of Dysport in Peroneus Longus in Equinus Foot Deformity in Children With Cerebral Palsy
Acronym: PerLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-52
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Equinus Foot Deformity in Children With Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A recent publication (Boulay et al. 2012) highlighted the role of the peroneus longus (PL) muscle in equinus foot deformity in children with hemiplegia. BoNT (Dysport) injections into this muscle have not yet been described in the literature. Based on the results of a previous study, the hypothesis is: this muscle may thus constitute a new therapeutic target for botulinum toxin injections in the early management of spastic equinus in children aged 2 years or older, before the onset of fixed neuro-orthopedic deformity and the midfoot break.

The aim of this retrospective study is to describe in intramuscular BoNT (Dysport) injections into PL based on the results obtained in a cohort of children (approximately 30 subjects) with cerebral palsy (hemiplegia or diplegia) and which have been treated in the service since 2007 until July 2012.

The investigators results are based on clinical, radiological and video evaluations. For this study, data will be collected in medical folder of each children belonging to this cohort.

All children (approximately 30 subjects) with cerebral palsy (hemiplegia or diplegia) which have been treated by BoNT (Dysport) intramuscular injections into PL in the service between 2007 and July 2012 will be screened. Subjects will be selected according to the following defined inclusion and exclusion criteria.

Data will be collected retrospectively (using a specific case report form designed for the study) in medical folder of each included subject for all visit of follow-up after BoNT (Dysport) injection into PL (since the first BoNT (Dysport) injection up to 2012). Then, data will be entered in a database. After that, they will be analysed .

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 6 years of age with cerebral palsy treated by intramuscular injection of BoNT (Dysport) into the PL (only) between 2007 and 2012.
* At least one BoNT (Dysport) injection performed into PL only
* Hemiplegic or diplegic subjects
* Dynamic equinus with hindfoot valgus with a documented premature onset activity of the peroneus longus which occurred earlier than the onset of Gastrocnemius Medialis (GM) activity, during terminal SW (i.e. EMG background data available).
* Evaluation based on Gross Motor Function Classification System (GMFCS ≤ 2) performed for children aged to 6-12 years (i.e available in the subject's medical folder).
* Feet Xrays data available before the first injection of BoNT (Dysport) and after for each subject
* Pre- and post-BoNT (Dysport) injection radiological data available in the subjects's medical folder

Exclusion Criteria:

* Equinus deformity due to a triceps surae contracture and a limb length discrepancy over 1 cm.
* Other muscle than PL injected with BoNT (Dysport) during the evaluation period (between the pre- ant post-BoNT (Dysport) radiological evaluation)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with cerebral palsy (hemiplegia or diplegia) which have been treated by BoNT (Dysport) intramuscular injections into PL in the service between 2007 and July 2012 .
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
foot morphology variation | 3 months
  radiological foot parameters including measured forefoot pronation (metatarsal stacking angle), midfoot planus (lateral talo-first metatarsal or Meary angle) and equinovalgus hind foot (incidence of postero-anterior ankle, calcaneal pitch and talocalcaneal angles)

SECONDARY OUTCOMES:
age | 3 months
  year
sex | 3 months
  female or male
weight | 3 months
Body Mass Index (BMI) | 3 months
Percentage of premature onset of muscle activity (EMG) | 3 months
Radiological data | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone, Marseille, France